CLINICAL TRIAL: NCT05260593
Title: Effectiveness of Phonophoresis With Vitamin B12 on Patients With Mild to Moderate Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Phonophoresis With Vitamin B12 on CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VB12CTS
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Vit. B12 Phonophoresis group) (Experimental): Patients in group (A) will receive phonophoresis with Vitamin B12. Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of vitamin B12 gel will be applied over the wrist. The following parameters will be used: intensity of 1.0 W/cm2 at a 1MHz frequency for 5 minutes and pulsed (25%) ultrasound waves to transfer the vitamin B12 gel. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.
  Interventions: Device: Vitamin B12 phonophoresis; Device: Wrist splint; Other: tendon and nerve gliding exercises
- Group B (Placebo-Phonophoresis with Vitamin B12) (Placebo Comparator): Patients in group (A) will receive placebo phonophoresis with Vitamin B12 gel. Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of Vitamin B12 gel will be applied over the wrist. The ultrasound probe will be held over the wrist using topical gel containing Vitamin B12 which was the same as in group A. Ultrasound device will seem to be working for 5 min period with light-off position. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.
  Interventions: Device: Placebo Vitamin B12 phonophoresis; Device: Wrist splint; Other: tendon and nerve gliding exercises

INTERVENTIONS:
Device: Vitamin B12 phonophoresis — Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of vitamin B12 gel will be applied over the wrist. The following parameters will be used: intensity of 1.0 W/cm2 at a 1MHz frequency for 5 minutes and pulsed (25%) ultrasound waves to transfer the vitamin B12 gel. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.
  Arms: Group A (Vit. B12 Phonophoresis group)
Device: Placebo Vitamin B12 phonophoresis — Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of Vitamin B12 will be applied over the wrist. The ultrasound probe will be held over the wrist using topical gel containing Vitamin B12 which was the same as in group A. Ultrasound device will seem to be working for 5 min period with light-off position. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.
  Arms: Group B (Placebo-Phonophoresis with Vitamin B12)
Device: Wrist splint — Patients were instructed to wear a neutral volar splint at night and while performing strenuous activities during the day for 5 weeks. Patients were given forms in order to check if they won't be compliant to the splint application and will be asked to bring the forms at the post treatment evaluation. Patients who won't check the form more than once a week will be regarded as non-compliant to splinting.
Other: tendon and nerve gliding exercises — During tendon-gliding exercises, the fingers will be placed in five discrete positions (straight, hook, fist, tabletop, and straight fist). During the median nerve-gliding exercise, six different hand and wrist positions will be used to mobilize the median nerve. During these exercises, the patient must maintain the neck and the shoulder in neutral position with a supinated forearm and elbow flexed 90 degrees. Each position must be maintained for 5 seconds. Each exercise will be repeated 10 times at each session and patients will be encouraged to apply exercise 3-5 times per day for 5 weeks.

SUMMARY:
The purpose of this study is to investigate efficacy of phonophoresis with vitamin B12 on median nerve distal latency, pain level and hand grip strength in patients with carpal tunnel syndrome. At least Fifty four Patients from both sexes will be recruited for this study from various hospitals in 6th October city

* Group A (n = 27): will receive Phonophoresis with Vitamin B12 gel.
* Group B (n = 27): will receive placebo phonophoresis with Vitamin B12 gel.

Median nerve distal latency, hand grip strength and numerical pain rating scale will be measured at baseline and after 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. at least Fifty Four patients with Mild to moderate CTS.
2. Age will range between 18 to 60 years old.
3. All patients will have Body mass index between 18.5 and 29.9 kg/m2.
4. Diagnosed by a physician according to American Association of Electrodiagnostic recent guidelines. (Jablecki et al., 2002).
5. A positive clinical provocative tests for CTS (Tinel test and Phalen test),
6. Patients with history of pain, paresthesia or numbness in the median nerve distribution, nocturnal pain, and night waking.

Exclusion Criteria:

1. Diabetic patients.
2. Hypertension patients.
3. Pregnant women
4. Cardiovascular patients
5. Patients with cervical spondylosis
6. Patients with cervical disc prolapse
7. Patients with Thoracic outlet syndrome
8. Patients with Carpal tunnel release surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-07-22 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Distal latency of median nerve sensory distal latency | Baseline and after 3 Weeks
  The Median sensory nerve (SNDL) distal latency was measured according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines with a Neuropack S1 MEB-9004 Nihon Koden (Japan). All measurements were performed in a room with the temperature kept at 25C.
Changes in Distal latency of median nerve motor distal latency | Baseline and after 3 Weeks
  The Median motor nerve (MNDL) distal latency was measured according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines with a Neuropack S1 MEB-9004 Nihon Koden (Japan). All measurements were performed in a room with the temperature kept at 25C.

SECONDARY OUTCOMES:
Changes in hand grip strength | Baseline and after 3 Weeks
  The hand grip strength (measured in Kilograms) was evaluated by the same investigator. Grip strength was tested by using Jamar hand held dynamometer following the American Society of Hand Therapists guidelines. The patient's arm was positioned with the shoulder adducted and neutrally rotated, the elbow was flexed at 90, the forearm and wrist were neutrally positioned while the participant was sitting. Patients were instructed to squeeze the handle as hard as they could, do maximal grip contraction for 2-5 s.
Changes in numeric pain rating scale (NPRS) | Baseline and after 3 Weeks
  An 11-point Numerical Pain Rating Scale (NPRS; 0 = no pain, 10 = maximum pain) was used to assess the patients' levels of hand pain pre and post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided